CLINICAL TRIAL: NCT03356392
Title: German Stroke Registry - Endovascular Treatment
Acronym: GSR-ET
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University Hospital of Cologne (Other); Klinikum rechts der Isar, Technical University of Munich (Unknown); RWTH Aachen University (Other); University Hospital Tuebingen (Other); Charite University, Berlin, Germany (Other); Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum (Unknown); Sana Klinikum Offenbach (Other); Goethe University (Other); Klinikum Dortmund (Unknown); KRH Klinikum Nordstadt (Unknown); Asklepios Klinik Altona (Unknown); Klinikum Altenburger Land (Unknown); Klinikum Stadt Hanau (Other); Klinikum Lüneburg (Unknown); Ludwig-Maximilians - University of Munich (Other); University of Göttingen (Other); Krankenhaus Buchholz (Unknown); Klinikum Osnabrück (Unknown); Wuerzburg University Hospital (Other); University of Giessen and Marburg (Unknown); Sana Kliniken Lübeck (Unknown); Mühlenkreiskliniken Minden (Unknown); radprax MVZ Nordrhein (Unknown); University Hospital Muenster (Other); University Medical Center Rostock (Other); Asklepios Klinik Wandsbek (Unknown); Elbe Kliniken (Unknown); Städtische Klinikum Braunschweig (Unknown); Allgemeines Krankenhaus Celle (Unknown); Bezirkskrankenhaus Günzburg (Unknown); Klinikum Bremen-Mitte, gGmbH (Other); University Medical Center Mainz (Other); Klinikum Köln-Merheim (Unknown); University Hospital, Bonn (Other)
Responsible Party: Sponsor
Other Study IDs: GSR-ET
Record Dates: First submitted 2017-11-22; First posted 2017-11-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke
Keywords: acute stroke, thrombectomy, endovascular treatment
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- stroke patients: acute stroke patients treated with endovascular treatment combined with or without
  Interventions: Other: telephone call d90

INTERVENTIONS:
Other: telephone call d90 — telephone call on day 90 to assess the primary outcome (mRs d90)

SUMMARY:
The German Stroke Registry (GSR) Endovascular Treatment is an academic, independent, prospective, multicentre, observational registry study. Consecutive patients treated with endovascular stroke treatment will be enrolled in German stroke centers. Patients receive regular care and data will be collected as part of clinical routine. Baseline clinical and procedural information as well clinical follow-up information during in-hospital stay, and up to 90 days of stroke onset are collected. Data collected include demographics, National Institute of Health Stroke Scale (NIHSS) on admission, pre-treatment ASPECTS, information on timing and success of interventional treatment, procedural complications, intracranial hemorrhage, and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke
* Eligible for intravenous thrombolysis (IVT) and IVT initiated within 4.5 hours after stroke onset
* Confirmed diagnosis of persistent occlusion of terminal carotid artery, middle cerebral artery (M1 or M2), or basilar artery consistent with symptoms
* Age >18 years
* Ethic approval in process

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all acute stroke patients with the clinical diagnosis of acute ischemic stroke, eligible for IVT and IVT initiated within 4.5 hours after stroke onset, Age >18 years
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
modified Ranking Scale (mRS) on day 90 | 90 days
  The scale is a commonly used measurement for the degree of disability or dependence in the daily activities of people who have suffered a stroke;
  scale range 0-6; with 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead. publication: van Swieten J, Koudstaal P, Visser M, Schouten H, et al. (1988). "Interobserver agreement for the assessment of handicap in stroke patients". Stroke. 19 (5): 604-607. doi:10.1161/01.str.19.5.604. PMID 3363593.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dichgans, Prof. Dr. med., Principal Investigator — LMU, Munich, Germany; Christian Gerloff, Prof. Dr. med., Principal Investigator — UKE, Hamburg, Germany
Locations (1):
- University Medical Center Hamburg-Eppendorf (UKE), Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deb-Chatterji M, Pinho J, Flottmann F, Meyer L, Broocks G, Brekenfeld C, Reich A, Fiehler J, Gerloff C, Thomalla G; GSR-ET Investigators. Health-related quality of life after thrombectomy in young-onset versus older stroke patients: a multicenter analysis. J Neurointerv Surg. 2022 Nov;14(11):1145-1150. doi: 10.1136/neurintsurg-2021-017991. Epub 2021 Dec 7. PMID 34876497
- [Background] Kniep H, Bechstein M, Broocks G, Brekenfeld C, Flottmann F, van Horn N, Geest V, Faizy TD, Deb-Chatterji M, Alegiani A, Thomalla G, Gellissen S, Fiehler J, Hanning U, Meyer L; German Stroke Registry-Endovascular Treatment (GSR-ET). Early surrogates of outcome after thrombectomy in posterior circulation stroke. Eur J Neurol. 2022 Nov;29(11):3296-3306. doi: 10.1111/ene.15519. Epub 2022 Aug 28. PMID 35933692
- [Derived] Hahn M, Groschel S, Lang LS, Othman AE, Groschel K, Uphaus T; German Stroke Registry - Endovascular Treatment (GSR-ET) investigators. Mortality within three months after nonfatal ischemic stroke treated by mechanical thrombectomy in routine care-data from the German Stroke Registry. Neurol Res Pract. 2025 Oct 1;7(1):71. doi: 10.1186/s42466-025-00427-7. PMID 41035079
- [Derived] Tong X, Jia B, Ma G, Zhang X, Fiehler J, Flottmann F, Bechstein M, Broocks G, Hanning U, Kniep HC, Thomalla G, Deb-Chatterji M, Schon G, Zhang Y, Gao F, Ma N, Mo D, Miao Z, Meyer L; as the ANGEL-ACT & GSR-ET study group. Relationship Between Thrombolysis-to-Puncture Time and Outcomes of Endovascular Thrombectomy in Acute Ischemic Stroke. Neurol Clin Pract. 2025 Aug;15(4):e200434. doi: 10.1212/CPJ.0000000000200434. Epub 2025 Jul 11. PMID 40656129
- [Derived] Heitkamp A, Hierholzer SM, Heitkamp C, Winkelmeier L, Meyer L, Bechstein M, Geest V, Broocks G, Brekenfeld C, Flottmann F, Schell M, Thomalla G, Faizy T, Fiehler J, Kniep HC, Gellissen S; German Stroke Registry -Endovascular Treatment (GSR-ET). Key to better outcomes in stroke intervention: early versus complete reperfusion in first pass recanalization. J Neurol. 2025 Jul 11;272(8):504. doi: 10.1007/s00415-025-13235-5. PMID 40646337
- [Derived] Single C, Mengel A, Laichinger K, Sartor-Pfeiffer J, Selo N, Hennersdorf F, Bender B, Deb-Chatterji M, Thomalla G, Mbroh J, Poli S, Ziemann U, Ernemann U, Feil K; German Stroke Registry-Endovascular Treatment (GSR). Sex-Related Differences in Outcomes of Endovascular Treatment in Large Vessel Occlusion Stroke-Analyses From the German Stroke Registry-Endovascular Treatment. Eur J Neurol. 2025 Mar;32(3):e70092. doi: 10.1111/ene.70092. PMID 40008680
- [Derived] Beckonert NM, Weller JM, Alegiani AC, Boeckh-Behrens T, Deb-Chatterji M, Hamann GF, Krause LU, Lehnen NC, Nitsch L, Poli S, Riedel C, Tiedt S, Zweynert S, Petzold GC, Dorn F, Bode FJ; GSR-ET investigators. Endovascular treatment of primary M3 occlusion stroke in clinical practice: analysis of the German Stroke Registry. Neurol Res Pract. 2024 Jul 18;6(1):36. doi: 10.1186/s42466-024-00330-7. PMID 39020409
- [Derived] Winkelmeier L, Heitkamp C, Faizy TD, Broocks G, Kniep H, Meyer L, Bester M, Brekenfeld C, Schell M, Hanning U, Thomalla G, Fiehler J, Flottmann F. Prognostic value of recanalization attempts in endovascular therapy for M2 segment middle cerebral artery occlusions. Int J Stroke. 2024 Apr;19(4):422-430. doi: 10.1177/17474930231214769. Epub 2023 Nov 22. PMID 37935652
- [Derived] Kniep H, Meyer L, Broocks G, Bechstein M, Guerreiro H, Winkelmeier L, Brekenfeld C, Flottmann F, Deb-Chatterji M, Alegiani A, Hanning U, Thomalla G, Fiehler J, Gellissen S; German Stroke Registry - Endovascular Treatment (GSR - ET). Predictors of functional outcome after thrombectomy for M2 occlusions: a large scale experience from clinical practice. Sci Rep. 2023 Oct 31;13(1):18740. doi: 10.1038/s41598-023-45232-x. PMID 37907482
- [Derived] Winkelmeier L, Faizy TD, Brekenfeld C, Heitkamp C, Broocks G, Bechstein M, Steffen P, Schell M, Gellissen S, Kniep H, Thomalla G, Fiehler J, Flottmann F; German Stroke Registry - Endovascular Treatment (GSR). Comparison of Thrombolysis In Cerebral Infarction (TICI) 2b and TICI 3 reperfusion in endovascular therapy for large ischemic anterior circulation strokes. J Neurointerv Surg. 2024 Oct 14;16(11):1076-1082. doi: 10.1136/jnis-2023-020724. PMID 37777256
- [Derived] Winkelmeier L, Faizy TD, Broocks G, Meyer L, Heitkamp C, Brekenfeld C, Thaler C, Steffen P, Schell M, Deb-Chatterji M, Hanning U, Kniep H, Maros ME, Thomalla G, Fiehler J, Flottmann FA; German Stroke Registry. Association Between Recanalization Attempts and Functional Outcome After Thrombectomy for Large Ischemic Stroke. Stroke. 2023 Sep;54(9):2304-2312. doi: 10.1161/STROKEAHA.123.042794. Epub 2023 Jul 26. PMID 37492970
- [Derived] Hahn M, Groschel S, Othman A, Brockstedt L, Civelek A, Brockmann MA, Groschel K, Uphaus T; German Stroke Registry Endovascular Treatment-Steering Committee. Real world data in mechanical thrombectomy: who are we losing to follow-up? J Neurointerv Surg. 2024 Apr 23;16(5):471-477. doi: 10.1136/jnis-2023-020435. PMID 37460214
- [Derived] Weller JM, Dorn F, Meissner JN, Stosser S, Beckonert NM, Nordsiek J, Kindler C, Riegler C, Keil F, Petzold GC, Bode FJ; GSR-ET investigators. Antithrombotic treatment and outcome after endovascular treatment and acute carotid artery stenting in stroke patients with atrial fibrillation. Neurol Res Pract. 2022 Sep 12;4(1):42. doi: 10.1186/s42466-022-00207-7. PMID 36089621
- [Derived] Weller JM, Dorn F, Meissner JN, Stosser S, Beckonert NM, Nordsiek J, Kindler C, Deb-Chatterji M, Petzold GC, Bode FJ; GSR-ET investigators. Endovascular thrombectomy in young patients with stroke. Int J Stroke. 2023 Apr;18(4):453-461. doi: 10.1177/17474930221119602. Epub 2022 Sep 7. PMID 35912650
- [Derived] Kniep H, Meyer L, Bechstein M, Broocks G, Guerreiro H, van Horn N, Brekenfeld C, Flottmann F, Deb-Chatterji M, Alegiani A, Thomalla G, Hanning U, Fiehler J, Gellissen S; GSR-ET (German Stroke Registry-Endovascular Treatment). How Much of the Thrombectomy Related Improvement in Functional Outcome Is Already Apparent at 24 Hours and at Hospital Discharge? Stroke. 2022 Sep;53(9):2828-2837. doi: 10.1161/STROKEAHA.121.037888. Epub 2022 May 13. PMID 35549377
- [Derived] Hahn M, Groschel S, Hayani E, Brockmann MA, Muthuraman M, Groschel K, Uphaus T; German Stroke Registry-Endovascular Treatment (GSR-ET) Study Group. Sex Disparities in Re-Employment in Stroke Patients With Large Vessel Occlusion Undergoing Mechanical Thrombectomy. Stroke. 2022 Aug;53(8):2528-2537. doi: 10.1161/STROKEAHA.121.037386. Epub 2022 Apr 21. PMID 35443786
- [Derived] Meyer L, Bechstein M, Bester M, Hanning U, Brekenfeld C, Flottmann F, Kniep H, van Horn N, Deb-Chatterji M, Thomalla G, Sporns P, Yeo LL, Tan BY, Gopinathan A, Kastrup A, Politi M, Papanagiotou P, Kemmling A, Fiehler J, Broocks G; German Stroke Registry-Endovascular Treatment (GSR-ET). Thrombectomy in Extensive Stroke May Not Be Beneficial and Is Associated With Increased Risk for Hemorrhage. Stroke. 2021 Oct;52(10):3109-3117. doi: 10.1161/STROKEAHA.120.033101. Epub 2021 Sep 2. PMID 34470489
- [Derived] Weller JM, Enkirch SJ, Bogs C, Braemswig TB, Deb-Chatterji M, Keil F, Kindler C, Maywald S, Schirmer MD, Stosser S, Solymosi L, Nolte CH, Bode FJ, Petzold GC; GSR-ET Investigators. Endovascular Treatment for Acute Stroke in Cerebral Amyloid Angiopathy. Stroke. 2021 Oct;52(10):e581-e585. doi: 10.1161/STROKEAHA.120.033014. Epub 2021 Aug 20. PMID 34412512
- [Derived] Maros ME, Brekenfeld C, Broocks G, Leischner H, McDonough R, Deb-Chatterji M, Alegiani A, Thomalla G, Fiehler J, Flottmann F; GSR Investigators*. Number of Retrieval Attempts Rather Than Procedure Time Is Associated With Risk of Symptomatic Intracranial Hemorrhage. Stroke. 2021 May;52(5):1580-1588. doi: 10.1161/STROKEAHA.120.031242. Epub 2021 Apr 5. PMID 33813864
- [Derived] Herm J, Schlemm L, Siebert E, Bohner G, Alegiani AC, Petzold GC, Pfeilschifter W, Tiedt S, Kellert L, Endres M, Nolte CH. How do treatment times impact on functional outcome in stroke patients undergoing thrombectomy in Germany? Results from the German Stroke Registry. Int J Stroke. 2021 Oct;16(8):953-961. doi: 10.1177/1747493020985260. Epub 2021 Jan 20. PMID 33472575
- [Derived] Flottmann F, Brekenfeld C, Broocks G, Leischner H, McDonough R, Faizy TD, Deb-Chatterji M, Alegiani A, Thomalla G, Mpotsaris A, Nolte CH, Fiehler J, Maros ME; GSR investigators*. Good Clinical Outcome Decreases With Number of Retrieval Attempts in Stroke Thrombectomy: Beyond the First-Pass Effect. Stroke. 2021 Jan;52(2):482-490. doi: 10.1161/STROKEAHA.120.029830. Epub 2021 Jan 20. PMID 33467875
- [Derived] Kupper C, Feil K, Wollenweber FA, Tiedt S, Herzberg M, Dorn F, Liebig T, Dieterich M, Kellert L; GSR investigators. Endovascular stroke treatment in orally anticoagulated patients: an analysis from the German Stroke Registry-Endovascular Treatment. J Neurol. 2021 May;268(5):1762-1769. doi: 10.1007/s00415-020-10369-6. Epub 2020 Dec 29. PMID 33373024
- [Derived] Ettelt P, Maier IL, Schnieder M, Bahr M, Behme D, Psychogios MN, Liman J; GSR-ET Collaborators. Bridging therapy is associated with improved cognitive function after large vessel occlusion stroke - an analysis of the German Stroke Registry. Neurol Res Pract. 2020 Jul 27;2:29. doi: 10.1186/s42466-020-00079-9. eCollection 2020. PMID 33324931
- [Derived] Wollenweber FA, Tiedt S, Alegiani A, Alber B, Bangard C, Berrouschot J, Bode FJ, Boeckh-Behrens T, Bohner G, Bormann A, Braun M, Dorn F, Eckert B, Flottmann F, Hamann GF, Henn KH, Herzberg M, Kastrup A, Kellert L, Kraemer C, Krause L, Lehm M, Liman J, Lowens S, Mpotsaris A, Papanagiotou P, Petersen M, Petzold GC, Pfeilschifter W, Psychogios MN, Reich A, von Rennenberg R, Rother J, Schafer JH, Siebert E, Siedow A, Solymosi L, Thonke S, Wagner M, Wunderlich S, Zweynert S, Nolte CH, Gerloff C, Thomalla G, Dichgans M, Fiehler J. Functional Outcome Following Stroke Thrombectomy in Clinical Practice. Stroke. 2019 Sep;50(9):2500-2506. doi: 10.1161/STROKEAHA.119.026005. Epub 2019 Jul 24. PMID 31337298
- [Derived] Alegiani AC, Dorn F, Herzberg M, Wollenweber FA, Kellert L, Siebert E, Nolte CH, von Rennenberg R, Hattingen E, Petzold GC, Bode FJ, Pfeilschifter W, Schafer JH, Wagner M, Rother J, Eckert B, Kraft P, Pham M, Boeckh-Behrens T, Wunderlich S, Bernkopf K, Reich A, Wiesmann M, Mpotsaris A, Psychogios M, Liman J, Maier I, Berrouschot J, Bormann A, Limmroth V, Spreer J, Petersen M, Krause L, Lowens S, Kraemer C, Zweynert S, Lange KS, Thonke S, Kastrup A, Papanagiotou P, Alber B, Braun M, Fiehler J, Gerloff C, Dichgans M, Thomalla G. Systematic evaluation of stroke thrombectomy in clinical practice: The German Stroke Registry Endovascular Treatment. Int J Stroke. 2019 Jun;14(4):372-380. doi: 10.1177/1747493018806199. Epub 2018 Oct 22. PMID 30346260
- See also: Homepage of German Stroke Registry — https://www.german-stroke-registry.de/german-stroke-registry